CLINICAL TRIAL: NCT06808854
Title: Variable-thread Versus Standard Dental Implants for Replacing Missing Teeth: a Randomized Controlled Trial
Brief Title: Variable-thread Versus Standard Dental Implants for Replacing Missing Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Momen Atieh, Professor and Chair (Periodontology), Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBRUMHS - 2024
Record Dates: First submitted 2025-01-07; First posted 2025-02-05 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-02

CONDITIONS: Dental Implants

STUDY DESIGN:
Intervention Model Description: Prospective, in which participants will be recruited and then followed up throughout a specified period of time.
  Randomized, parallel designed, concurrent controlled trial with participants randomly allocated to either test or control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Variable-thread implants (Experimental): The placement of a variable-thread implant to replace single missing posterior tooth
  Interventions: Procedure: Dental implant treatment (variable-thread implants)
- Standard implants (Active Comparator): The placement of standard implant to replace single missing posterior tooth
  Interventions: Procedure: Dental implant treatment (standard implants)

INTERVENTIONS:
Procedure: Dental implant treatment (variable-thread implants) — Replacement of a missing tooth with a dental implant with variable-thread implants
  Arms: Variable-thread implants
Procedure: Dental implant treatment (standard implants) — Replacement of a missing tooth with a dental implant with standard implants
  Arms: Standard implants

SUMMARY:
Background and objectives:

Primary and secondary implant stability remain the most relevant and reliable clinical indicator for long-term survival of dental implants. Hence modifications of surface characteristics and implant macro-designs were introduced over the last two decades to enhance osseointegration during the initial phase of healing. In this context, a variable-thread self-cutting implant design was recently introduced to improve primary stability. At present, there are limited number of studies that evaluated this variable-thread implant design. These studies were mostly experimental, of short duration and limited number of participants. Therefore, the aim of the present randomized controlled trial is to compare two implant designs (variable-thread versus standard) in terms of clinical, radiographic and patient-reported outcomes.

Methods:

A total of 24 participants, who require replacement of a posterior single tooth with dental implant, will be randomly allocated to two equal sized groups. In the test group, the participants will receive variable-thread implants, while standard implants will be placed to replace missing teeth in the control group. In addition to evaluating implant stability, the trial will also report on clinical and radiographic implant outcomes at various time points.

DETAILED DESCRIPTION:
Introduction

Implant stability is a prerequisite for successful osseointegration and implant survival as implant micro-motion can compromise osseointegration and lead to implant failure. Maintenance of implant stability over time has been considered one of the implant success criteria that is identified at the primary or secondary level. Primary implant stability occurs as a result of bone compression and mechanical interlocking between implant surface and bone at the time of implant placement. Therefore, primary stability can be largely influenced by implant surface characteristics and implant design in terms of microstructure, thread design and geometry as well as bone quality and quantity. In contrast, secondary implant stability is a biologically mediated process by which bone matures and remodels at the bone-implant interface.

Primary and secondary implant stability remain the most relevant and reliable clinical indicator for long-term survival of dental implants. Hence modifications of surface characteristics and implant macro-designs were introduced over the last two decades to enhance osseointegration during the initial phase of healing. In this context, an implant design was recently introduced to improve primary stability particularly in areas of poor bone quality such as the posterior maxilla. The recently introduced implant has self-cutting self-drilling body with variable thread configurations that are designed to allow controlled compaction and condensation of bone during insertion thus enhancing the initial bone to implant contact. It is claimed that high primary stability is achieved by a controlled bone compaction and densification mechanism resulting from the double variable thread design and the apical sharp threads. In addition, the implant is made up of titanium-zirconium alloy that provide strength, high resistance to loading and biocompatibility. Its moderately rough hydrophilic sandblasted and acid-etched (SLActive) surface can also improve bone-implant contact during the early phase of osseointegration.

At present, there are limited number of studies that evaluated this variable-thread implant design. These studies were mostly experimental, of short duration and limited number of participants. Therefore, the aim of the present randomized controlled trial is to compare two implant designs (variable-thread versus standard) in terms of clinical, radiographic and patient-reported outcomes.

Objectives:

The aims of the present randomized controlled trial are:

* To evaluate implant stability.
* To evaluate the changes in peri-implant marginal bone level.
* To evaluate implant survival rates.
* To evaluate biological and technical complications during the follow-up period.

ELIGIBILITY:
Inclusion criteria

* Aged more than 18 years.
* Good general health (ASA I or II, according to the American Academy of Anesthesiology).
* Require replacement of a posterior single missing tooth with a dental implant.
* Controlled oral hygiene (full-mouth plaque and bleeding scores ≤ 25% at baseline.
* Good compliance and commitment to attend follow-up review appointments.
* Willing to provide informed consent. Exclusion criteria
* A healing period of less than four months postextraction at implant site.
* Localized/generalized periodontitis.
* Bone metabolic disease and/or taking medications that affect bone metabolism.
* Long term use of non-steroidal anti-inflammatory medications.
* History of malignancy, radiotherapy or chemotherapy.
* Pregnant or lactating women.
* Severe bruxism or parafunctional habits.
* Large occlusal discrepancies.
* Smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Implant stability measurements | "during implant placement procedure" "1 year" "up to 24 weeks" "through study completion, an average of 1 year".
  A resonance frequency analysis device will used to measure the stability of the dental implant. The measurements will be recorded The use of a resonance frequency analysis device involves the following steps: attach the sensor to the implant, activate the device to measure resonance frequency, read the implant stability quotient (ISQ) value displayed on the device.

SECONDARY OUTCOMES:
Changes in peri-implant marginal bone level | "during implant placement procedure" "1 year" "up to 24 weeks" "through study completion, an average of 1 year".
  Changes in peri-implant marginal bone level will be assessed using standardized peri-apical radiograph
Implant survival rate | "1 year" "up to 24 weeks" "through study completion, an average of 1 year".
  Implant survival rate will be assessed clinically after one year of implant restoration and annually up to three years. Unlike other measurements, implant survival, defined as a dental implant that remains in place and functional, will be only assessed once a year.
Biological and technical complications | "1 year" "up to 24 weeks" "through study completion, an average of 1 year".
  Biological and technical complications will be recorded during the follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- MBRU, Dubai, United Arab Emirates